CLINICAL TRIAL: NCT02306200
Title: Cardiovascular Health Improvement Project
Acronym: CHIP
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Marion Hofmann Bowman, Associate Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00052866
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Aortic Aneurysm; Aortic Dissection; Bicuspid Aortic Valve (BAV); Heart Failure; Cardiovascular Diseases
Keywords: Aorta; Abdominal Aortic Aneurysm (AAA); Thoracic Aortic Aneurysm (TAA); Bicuspid Aortic Valve (BAV); Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Bicuspid Aortic Valve Disease; Heart Failure; Cardiovascular Diseases; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Biospecimen Retention: Samples With DNA — Blood, Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aortic Disease: Patients with a diagnosis of any form of Aortic Disease
- Controls: Patients without a diagnosis of Aortic Disease

SUMMARY:
The goal of this project is to establish a biobank of clinical information, DNA, plasma, and aortic tissue samples from patients with cardiovascular disease as well as healthy controls.

DETAILED DESCRIPTION:
The goal of this project is to establish a biobank of clinical information, DNA, plasma, and aortic tissue samples from patients with cardiovascular disease as well as healthy controls. The aims of the study are to collect biological specimens (blood, plasma, serum, aortic tissue) and family history; establish a biobank, establish a comprehensive database with information from consented patients, and provide researchers with high quality well annotated DNA samples with demographic and clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 who is able/willing to give informed consent
* Patients <18 years of age with parental consent and assent (if assent is applicable for their age)
* Diagnosis of:
* aortic pathology potentially due to a known or suspected inherited condition
* Idiopathic aortic aneurysm
* Interesting of novel vascular pathology in the aorta or main branches
* Family history of aortic or vascular disease
* Other cardiovascular disease
* Healthy controls with no apparent cardiovascular disease

Exclusion Criteria:

- Not willing or able to sign the consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2013-08; Primary Completion 2053-08 (Estimated); Study Completion 2053-08 (Estimated)

PRIMARY OUTCOMES:
Establishing a biobank of patients with Aortic Disease | 40 years
  Establish a biobank of blood, serum, plasma, tissue, and clinical data of patients with any form of aortic disease

CONTACTS AND LOCATIONS:
Overall Officials: Marion A Hofmann Bowman, PhD, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Love-Nichols J, Uhlmann WR, Arscott P, Willer C, Hornsby W, Roberts JS. A survey of aortic disease biorepository participants' preferences for return of research genetic results. J Genet Couns. 2021 Jun;30(3):645-655. doi: 10.1002/jgc4.1341. Epub 2020 Dec 14. PMID 33319384